CLINICAL TRIAL: NCT06234709
Title: Comorbidity With Greatest Impact on Mortality Considering Different Admission Diagnosis and After Landmark Time in an Intensive Care Population Compared to the General Population
Brief Title: Long-term Mortality After Intensive Care Considering Comorbidity and Admission Diagnoses
Status: Completed | Type: Observational
Sponsor: Anna Aronsson (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor-Investigator, Anna Aronsson, Principal Investigator, Uppsala University
Organization: Uppsala University (Other)
Other Study IDs: Anna Aronsson Dannewitz
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Critical Care
Keywords: Comorbidity; Intensive care; SAPS3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a register-based study

The aim of this study is to investigate how common comorbidity is in different age groups and which comorbidity that has the greatest impact on mortality considering different admission diagnosis and after the acute phase compared to the general population. Also, how different degrees of comorbidity affect mortality, adjusted for other comorbidities and SAPS 3?

DETAILED DESCRIPTION:
The study population included all patients > 16 years old admitted to an ICU during the years 2006 to 2012 and registered in the Swedish Intensive Care Registry (SIR).

Hospital discharge diagnoses from in-patient care five years preceding the index time for the ICU admission were extracted from the National Patient Register (NPR) and linked to ICU admissions using unique person identity numbers. Follow-up for all-cause mortality were extracted from the cause of death register at NPR.

ELIGIBILITY:
Inclusion Criteria:

The study population included all patients > 16 years old admitted to an ICU during the years 2006 to 2012 and registered in the Swedish Intensive Care Registry (SIR)

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population included all patients > 16 years old admitted to an ICU during the years 2006 to 2012 and registered in the Swedish Intensive Care Registry (SIR)
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | january 1, 2005 til december 31, 2016
  Extracted from the cause of death register at National Patient Registry in Sweden.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Aronsson Dannewitz, med mag, Principal Investigator — Uppsala university department of surgical sciense
Locations (1):
- Uppsala university department of surgical sciences, Uppsala, Sweden

REFERENCES:
- [Derived] Aronsson Dannewitz A, Svennblad B, Michaelsson K, Lipcsey M, Gedeborg R. The long-term conditional mortality rate in older ICU patients compared to the general population. Crit Care. 2024 Nov 14;28(1):368. doi: 10.1186/s13054-024-05147-z. PMID 39543756